CLINICAL TRIAL: NCT03594305
Title: From Obstacles to Opportunities for Family Planning in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Fuller Theological Seminary (Unknown); St. Paul College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1605017246
Record Dates: First submitted 2018-06-05; First posted 2018-07-20 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial in which villages are randomized to receive or not to receive the intervention.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Intervention Arm (Experimental): Villages randomized to this arm will receive a one-day educational seminar, which their religious leaders of all denominations will be invited to attend. The seminar will address religious, cultural, and medical aspects of family planning. Leaders who attend will also have the opportunity to participate in mentorship group discussions after the intervention. In addition, both villages will have standard teaching provided by nurses at dispensaries about family planning, and a continual supply of contraceptive options at dispensaries in all villages will be ensured.
  Interventions: Behavioral: Educational seminar
- Control arm (No Intervention): Villages randomized to this arm will not receive the educational seminar. These villages will have standard teaching provided by nurses at dispensaries about family planning, and a continual supply of contraceptive options at dispensaries in all villages will be ensured.

INTERVENTIONS:
Behavioral: Educational seminar — Religious leaders will be invited to participate in a one-day seminar led by Tanzanian religious leaders and physicians. The religious, cultural, and medical aspects of family planning will be discussed and seminar attendees will be given ample time for group discussions.
  Arms: Educational Intervention Arm

SUMMARY:
The investigators will conduct a cluster randomized trial to determine the effectiveness of an educational intervention for religious leaders in promoting uptake of family planning in Tanzania.

DETAILED DESCRIPTION:
In this community randomized trial, the investigators will randomize 12 rural villages to receive an educational seminar for their religious leaders about family planning. The investigators will compare these uptake of family planning in these 12 villages with 12 matched villages whose religious leaders do not attend an educational seminar about family planning. The investigators will also determine women's reasons for seeking family planning at the village dispensaries..

Prior to the start of the trial, the study team will ensure that dispensaries in all villages in the trial will have a reliable supply of contraceptive options. To mitigate the effect of economic barriers and medication shortages on access to contraception, a dedicated medication supply team will make certain that all dispensaries remain well-stocked with standard contraceptives that are free from the Tanzanian Ministry of Health. These include oral contraceptive pills, implants, injections, copper intrauterine devices, and condoms.

Villages will be paired by proximity (within 50 kilometers of one another). Within the pair, one village will be randomly assigned, using a computer-generated algorithm, to receive the intervention of religiously- and culturally-informed teaching intervention about family planning for religious leaders. The other village will be the control village. Each intervention village will be followed, and its religious leaders mentored in groups, for 12 months after the start of the intervention. Mentorship groups of 25 leaders, led by the study team, will meet for 1 hour per month. The investigators will also conduct focus groups in both intervention and control villages to understand community perceptions of family planning.

ELIGIBILITY:
Inclusion Criteria:

* Rural villages in northwest Tanzania with populations between 8,000 and 20,000
* Village dispensaries present to measure uptake of family planning
* Located in close proximity (50 km or less) to another eligible village with which it can be paired

Exclusion Criteria:

* Private dispensaries at which family planning uptake would be missed

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Uptake of family planning at village dispensaries | 12 months
  The investigators will measure the percent of the population seeking modern contraception.

SECONDARY OUTCOMES:
Pregnancy rates | 12 months
  The investigators will obtain pregnancy rates for the village stratified by age.
Reasons for seeking family planning | 12 months
  Women seeking family planning will answer a short structured yes/no questionnaire to determine the sources from which they were encouraged to seek family planning.
Couple-years of protection | 12 months
  The investigators will use the types of family planning accessed to calculate couple-years of protection per given population number, according to conversion numbers provided by USAID (https://www.usaid.gov/what-we-do/global-health/family-planning/couple-years-protection-cyp)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Downs, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- St. Paul College, Mwanza, Tanzania

REFERENCES:
- [Derived] Mwakisole AH, Lambert VJ, Nzali A, Aristide C, Laizer E, Cordeiro AA, Gregory L, Mwakisole N, Nicol CEW, Paul N, Kalluvya SE, Kihunrwa A, Downs DJ, Wamoyi J, Downs JA, Lee MH. Partnerships with religious leaders to promote family planning in rural Tanzania: an open-label, cluster randomised trial. Lancet Glob Health. 2023 Dec;11(12):e1943-e1954. doi: 10.1016/S2214-109X(23)00453-9. PMID 37973342